CLINICAL TRIAL: NCT04738162
Title: Clinical Safety Study on 5-Aminolevulinic Acid (5-ALA) in Children and Adolescents With Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universität Münster (Other)
Collaborators: photonamic GmbH & Co. KG (Industry); medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UKM2013_0034; 2014-005669-54 (EudraCT Number)
Record Dates: First submitted 2020-05-13; First posted 2021-02-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor, Pediatric
Keywords: 5-ALA; intra-axial; Fluorescence-guided resection; pediatric
MeSH Terms: conditions — Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5-Aminolevulinic Acid (5-ALA) (Experimental): Application of 5-ALA oral solution followed by fluorescence-guided brain tumor resection
  Interventions: Drug: 5-Aminolevulinic Acid Hydrochloride, Oral

INTERVENTIONS:
Drug: 5-Aminolevulinic Acid Hydrochloride, Oral — Application of 5-ALA oral solution (20mg/kg bw) 4 hours (range 3.5-4.5 hours) prior to anesthesia followed by fluorescence-guided tumor resection Tumor resection is performed conventionally using a surgical microscope. A change from white light to blue light is possible at anytime to make the fluorescence visible
  Other Names: Gliolan

SUMMARY:
In this prospective, open, single-armed, multicenter, phase II study for application of 5-ALA in children and adolescents with brain tumors 80 patients will be investigated.

Primary objective of the study is to determine the safety of 5-ALA for fluorescence-guided resections in children and adolescents with intra-axial brain tumors.

Secondary objectives are

* to determine whether fluorescent tissue truly signifies tumor (positive predictive value) in various pediatric brain tumors
* to determine the degree of tumor resection on early post-operative MRI
* and to determine the pharmacokinetics of 5-ALA in this population.

DETAILED DESCRIPTION:
In 2007, 5-aminolevulinic acid (5-ALA) was approved in Europe by the European Medicines Agency (EMA) (brand name: Gliolan®) for "the visualization of malignant tissue during surgery for malignant glioma (WHO III and IV) in adults." Similarly, approval for 5-ALA was granted by the FDA in 2017 as an "optical imaging agent indicated in patients with gliomas (suspected World Health Organization Grades III or IV on preoperative imaging) as an adjunct for the visualization of malignant tissue during surgery" (brand name: Gliolan®). Goal of the study is to investigate if the use of 5-ALA is safe in children and get preliminary information on the type of paediatric brain tumors which are suitable for fluorescence-guided resection with 5-ALA.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 - <18 years
* First radiological diagnosis of intra-axial, contrast-enhancing tumor on MRI or recurrent supratentorial intra-axial brain tumor (malignant glioma, astrocytoma, malignant ependymoma, atypical teratoid rhabdoid tumors (AT/RT), Oligodendroglioma, etc.)
* Resection is part of therapeutic strategy with an emphasis on neurological safety
* Informed consent by the parents or guardians and if possible assent of the patient after education of purpose and risks of study. Patients that are able to understand should provide assent to participate in the trial
* Female adolescents: not pregnant (pregnancy test required for adolescents of child-bearing age) and not breast-feeding (for at least 24 hours after Gliolan intake). Female patients of childbearing potential and male patients who are sexually active must be practising a highly effective method of birth control up to 6 weeks after the tumor operation consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials.

Exclusion Criteria:

* Extra-axial tumors such as craniopharyngioma
* Entities precluding surgical resection
* Acute or chronic porphyria
* Hypersensitivity to 5-ALA or porphyrins
* Renal insufficiency: serum creatinine > 2x upper limit of normal (ULN)
* Hepatic insufficiency: serum bilirubin > 2x ULN, serum γ-glutamyl transferase > 2,5 x ULN, alanine transaminase (ALT) and aspartate transaminase (AST)> 2,5 ULN
* Blood clotting: INR (international normalized ratio) out of acceptable limits
* Other malignant disease
* Patients with pre-existing cardiovascular diseases
* Co-administration with other potentially phototoxic substances (e.g. tetracyclines, sulfonamides, fluoroquinolones, hypericin extracts)
* Planned administration of potentially hepatotoxic substances within 24 hours after 5-ALA administration

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Safety of 5-ALA for fluorescence-guided resections in children and adolescents determined as incidence of adverse events of CTCAE grade III-V. | up to 6 weeks after tumor resection
  Incidence of adverse events of CTCAE grade III, IV or V (excluding chemotherapy-associated toxicities) during and after 5-ALA fluorescence-guided resections in children and adolescents

SECONDARY OUTCOMES:
True positive rate of fluorescence for indicating tumor | Day 0: during the surgery
  Biopsies will be taken during tumor resection. The true positive rate of 5 ALA induced fluorescence for three different tumor regions, i.e. the number of fluorescing tumor samples containing tumor cells divided by the number of all tumor samples from 1) the tumor bulk, 2) the border area and 3) the suspected infiltration zone. A stratification will be performed depending on whether surgery is for newly diagnosed or recurrent tumor.
Determination of the percentage of patients with gros total resection and subtotal resection | up to 72h after surgery
  For every patient in whom a complete resection of enhancing tumor is expected a priori, it will be assessed whether there is residual contrast-enhancement or not on early post-operative MRI. The volume of contrast-enhancing tumor on early post-operative MRI (up to 72h after surgery) in cm3 will be determined. If the volume is < 0.175cm3, the patient will be classified as "gros total resection". If the volume is >0.175cm3, the patient will be classified as "subtotal resection". Percentage of patients for both groups will be determined.
Correlation of residual contrast-enhancing tumor with residual fluorescence after surgery | Day 0: during the surgery
  For both groups (patients with gros total and subtotal resection) the percentage of patients with residual fluorescence at end of surgery, as determined during the surgery by the operating surgeon (yes/no), will be calculated.
Determination of protoporphyrin IX (PPIX) in serum to analyse AUC (Area under the curve) of PPIX | 3-6 hours, 6-9 hours and 9-12 hours after surgery
  The investigators aim to determine 5-ALA pharmacokinetics in children and adolescents from PPIX plasma levels in order to assess if the pharmacokinetics differ between adults and children. Pharmacokinetic data will be analyzed using population pharmacokinetic software approach using nonlinear-mixed effects modelling (NONMEM). In order to assess if the pharmacokinetics are similar, the area under the curve (AUC) for PPIX as a measure of 5-ALA exposure will be calculated. For this purpose protoporphyrin IX will be measured in serum 3 times within 12h after 5-ALA-administration.
Determination of protoporphyrin IX (PPIX) in serum to determine interpolated maximum plasma concentration (Cmax) of PPIX. | 3-6 hours, 6-9 hours and 9-12 hours after surgery
  Protoporphyrin IX will be measured in serum 3 times within 12h after 5-ALA-administration. Pharmacokinetic data will be analyzed using population pharmacokinetic software approach using nonlinear-mixed effects modelling (NONMEM). Using the model, interpolated maximum plasma concentration (Cmax) of PPIX will be determined for every patient.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stummer, Prof., Principal Investigator — University Hospital Muenster
Locations (7):
- Germany (6):
  - Universitätsklinikum Augsburg, Klinik für Neurochirurgie, Augsburg
  - Universitätsklinikum Essen, Klinik für Neurochirurgie, Essen
  - Universitätsmedizin Mainz, Klinik und Poliklinik für Neurochirurgie, Mainz
  - Neurochirurgische Klinik der Universität München (LMU), München
  - University Hospital Münster, Klinik für Neurochirurgie, Münster
  - Universitätsklinikum Tübingen, Klinik für Neurochirurgie, Tübingen
- Prinses Máxima Centrum voor kinderoncologie BV, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No